CLINICAL TRIAL: NCT00473499
Title: Paclitaxel-Eluting PTCA-Balloon in Combination With the Coroflex Blue Stent vs the Sirolimus Coated Cypher Stent in the Treatment of Advanced Coronary Artery Disease - Substudy Homburg/Saar
Brief Title: PEPCAD III Substudy: Stem Cell Mobilization
Acronym: PEPCADIIIsub
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital, Saarland (Other)
Responsible Party: Prof. Dr. Bruno Scheller, University Hospital, Saarland
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BBM-VS54-HOM
Record Dates: First submitted 2007-05-14; First posted 2007-05-15 (Estimated); Last update posted 2010-06-30 (Estimated); Status verified 2010-06

CONDITIONS: Coronary Artery Disease
Keywords: drug eluting balloon; drug eluting stent; stem cells
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- DEBlue stent (Experimental): Paclitaxel coated balloon with CoCr stent mounted on it
  Interventions: Device: DEBlue vs Cypher vs BMS
- Cypher stent (Active Comparator)
  Interventions: Device: DEBlue vs Cypher vs BMS
- Coroflex Blue stent (Placebo Comparator)
  Interventions: Device: DEBlue vs Cypher vs BMS

INTERVENTIONS:
Device: DEBlue vs Cypher vs BMS — BMS vs DES vs DEB+BMS

SUMMARY:
The aim of the PEPCAD III substudy is to assess the efficacy of the Paclitaxel-eluting DEBlue stent system in the treatment of stenoses in native coronary arteries compared to the Sirolimus-eluting Cypher stent by intravascular ultrasound (IVUS) and to study the influence of both devices on endothelial function, coronary flow reserve, and stem cell mobilization.

DETAILED DESCRIPTION:
The aim of the PEPCAD III substudy is to assess the efficacy of the DEBlue® Paclitaxel-eluting stent system in the treatment of stenoses in native coronary arteries compared to the Sirolimus-eluting Cypher stent by intravascular ultrasound (IVUS) and to study the influence of both devices on endothelial function, coronary flow reserve, and stem cell mobilization. This study is a prospective, randomized, single-center, two-armed phase-II study. During the PEPCAD III trial, 40 patients of the Homburg / Saar center will be randomly assigned to ei-ther one of the treatment groups (20 patients treated with DEBlue, 20 patients with Cypher®). Patients with stable or selected forms of unstable angina or documented ischemia due to a significant lesion in a native coronary artery will be included. Vessels may not supply an en-tirely infarcted myocardial area. Additional 20 patients receiving uncoated stents (Coroflex® Blue, B.Braun) will undergo the same diagnostic procedures.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stable or unstable angina or documented ischemia due to a significant lesion in a native coronary artery
* Patients eligible for coronary revascularization by means of PCI
* Intention to treat one lesion with one stent
* Patients suitable for coronary revascularization of any sort (balloon angioplasty, device-assisted balloon-angioplasty, or coronary artery bypass grafting)
* Patients must be ≥ 18 years of age
* Women of childbearing potential may not be pregnant nor have the desire to becoming pregnant during the first year following the study procedure. Hence, patients will be advised to use an adequate birth control method up to and including 9 months follow-up
* Patients who are mentally and linguistically able to understand the aim of the study and to show sufficient compliance in following the study protocol
* Patients must agree to undergo the 9 months angiographic follow-up
* Patients must agree to undergo the 1 and 3 year clinical follow-up
* Patient is able to verbally acknowledge an understanding of the associated risks, benefits, and treatment alternatives to therapeutic options of this trial, e.g. balloon angioplasty by means of the Paclitaxel-eluting PTCA-balloon catheter in combination with the Coroflex BlueTM stent or the Sirolimus-eluting CypherTM stent. The patients, by providing informed consent, agree to these risks and benefits as stated in the patient informed consent document.
* Significant stenoses in native coronary arteries with nominal stent diameters between ≥ 2.5 mm and ≤ 3.5 mm and < 24 mm in length

Exclusion Criteria:

* Unprotected left main
* In stent restenosis
* Indication for more than one lesion to treat, even as staged procedure
* Intended bifurcational stenting
* Patients requiring chronic anticoagulation
* SVG and AG
* Acute MI (STEMI, NSTEMI)
* Cardiogenic shock
* Chronic total occlusions
* Pregnancy
* Patients with stand alone balloon angioplasty, or stent deployment 6 months prior to enrolment into this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2007-07; Primary Completion 2009-03 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
stem cell mobilization and differentiation | 7 days
endothelial function | 9 months

SECONDARY OUTCOMES:
late lumen loss | 9 months
MACE | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Scheller, Principal Investigator — Klinik fuer Innere Medizin III, Universitaetsklinikum des Saarlandes, Homburg/Saar, Germany
Locations (1):
- Klinik fuer Innere Medizin III, Universitaetsklinikum des Saarlandes, Homburg / Saar, Saarland, Germany

REFERENCES:
- [Background] Scheller B, Speck U, Bohm M. Prevention of restenosis: is angioplasty the answer? Heart. 2007 May;93(5):539-41. doi: 10.1136/hrt.2007.118059. PMID 17435062
- [Background] Scheller B, Hehrlein C, Bocksch W, Rutsch W, Haghi D, Dietz U, Bohm M, Speck U. Treatment of coronary in-stent restenosis with a paclitaxel-coated balloon catheter. N Engl J Med. 2006 Nov 16;355(20):2113-24. doi: 10.1056/NEJMoa061254. Epub 2006 Nov 13. PMID 17101615
- [Background] Speck U, Scheller B, Abramjuk C, Breitwieser C, Dobberstein J, Boehm M, Hamm B. Neointima inhibition: comparison of effectiveness of non-stent-based local drug delivery and a drug-eluting stent in porcine coronary arteries. Radiology. 2006 Aug;240(2):411-8. doi: 10.1148/radiol.2402051248. PMID 16864669
- [Background] Scheller B, Speck U, Abramjuk C, Bernhardt U, Bohm M, Nickenig G. Paclitaxel balloon coating, a novel method for prevention and therapy of restenosis. Circulation. 2004 Aug 17;110(7):810-4. doi: 10.1161/01.CIR.0000138929.71660.E0. Epub 2004 Aug 9. PMID 15302790
- [Background] Inoue T, Sata M, Hikichi Y, Sohma R, Fukuda D, Uchida T, Shimizu M, Komoda H, Node K. Mobilization of CD34-positive bone marrow-derived cells after coronary stent implantation: impact on restenosis. Circulation. 2007 Feb 6;115(5):553-61. doi: 10.1161/CIRCULATIONAHA.106.621714. Epub 2007 Jan 29. PMID 17261663
- [Derived] Clever YP, Cremers B, Speck U, Dietz U, Bohm M, Scheller B. Influence of a paclitaxel coated balloon in combination with a bare metal stent on restenosis and endothelial function: comparison with a drug eluting stent and a bare metal stent. Catheter Cardiovasc Interv. 2014 Aug 1;84(2):323-31. doi: 10.1002/ccd.25184. Epub 2013 Sep 30. PMID 23996969